CLINICAL TRIAL: NCT06362213
Title: Gaining Insight Into Dual Sensory Loss: Quantitative Study
Brief Title: Gaining Insight Into Dual Sensory Loss
Acronym: DSL
Status: Not yet recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Royal Dutch Visio (Other)
Responsible Party: Principal Investigator, R.M.A. (Ruth) van Nispen, prof.dr. R.M.A. van Nispen, Amsterdam UMC, location VUmc
Other Study IDs: NL76924.029.22
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Dual Sensory Impairment of Vision and Hearing
Keywords: information access; mobility; communication; fatigue; visual acuity; contrast sensitivity; visual field; hearing threshold; speech understanding in noise; speech understanding in silence; directional hearing
MeSH Terms: conditions — Communication; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- participants with dual sensory loss: participants with both vision and hearing loss
- participants with vision loss: participants with vision loss only
- participants with hearing loss: participants with hearing loss only
- participants with normal vision and hearing: participants without vision or hearing loss

SUMMARY:
The goal of this observational study is to explore difficulties in information access, mobility, communication and fatigue in people with combined vision and hearing impairments. The main question it aims to answer is:

• What influence do varying severities of vision and hearing loss have on information access, mobility, communication and fatigue.

Participants will fill out questionnaires and the researchers will measure their vision and hearing functions.

DETAILED DESCRIPTION:
People with dual sensory loss have impairments in both vision and hearing. When the impairments are severe, it will become more difficult to compensate for these impairments. This can result in difficulties, for example in the areas of access to information, communication, fatigue and/or mobility. Now, we do not know which problems arise from different combinations and levels of impairments in visual acuity, contrast sensitivity, visual field, hearing threshold, directional hearing and speech understanding. We also do not know how this influences the areas of access to information, communication, fatigue and mobility.

The objective of this study is to determine which problems arise from different levels of impairments in visual and auditory functions. We will especially focus on the areas of access to information, communication, fatigue and mobility.

Study design

Participants' visual (visual acuity, visual field, contrast sensitivity) and auditory functions (hearing threshold, directional hearing, speech understanding) will be measured. We will use the following materials:

* ETDRS card
* Vistech card
* Octopus perimeter
* Affinity compact audiometer
* 8 Genelec 8020 DPM speakers (to measure directional hearing)
* Digits in Noise (DIN) test and NVA word lists

Several questionnaires will be filled out to measure difficulties in the areas of access to information, communication, fatigue and mobility:

* Dutch ICF Activity Inventory - domains watching TV, using a computer, using a telephone, mobility outdoors (walking), using public transportation and feeling fit
* Speech, Spatial and Qualities of Hearing Scale
* Spatial Localization Questionnaire
* Fatigue Assessment Scale

Study population:

* 150 people with dual sensory loss
* 50 people with a visual impairment
* 50 people with an auditory impairment
* 50 people with normal vision and hearing

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Good understanding of the Dutch language
* Clients: visual and/or auditory impairment (congenital or acquired)
* Other participants: normal vision and hearing

Exclusion Criteria:

* Impaired cognitive functioning

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with dual sensory loss have impairments in both vision and hearing, which can range from total vision and hearing loss to having limited residual vision and hearing.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
information access | 1 day
  Access to information will be measured with the Dutch ICF Activity Inventory (subscales 'Watching TV', 'Using a computer' and 'Using a telephone'). These subscales consist of 11, 13 and 5 items, respectively (29 items in total). All items are scored on a 5-point likert scale.
mobility | 1 day
  Mobility will be measured with the Dutch ICF Activity Inventory (subscales 'Mobility outdoors (walking)' and 'Using public transportation'). These subscales consist of 16 and 15 items, respectively (31 items in total). All items are scored on a 5-point likert scale. Secondly, the Spatial Localization Questionnaire20 will be used, consisting of 35 items, describing common scenarios. The following question structure is provided under each of the scenarios:
  Can you complete this task solely with your current vision? If yes, how difficult is it? (rated on a 5-point likert scale) Can you complete this task solely with your current hearing? If yes, how difficult is it? (rated on a 5-point likert scale) Would you primarily rely on your vision or hearing for this task? Do you use the other sense for this task at all?
communication | 1 day
  Communication will be measured with the Speech, Spatial and Qualities of Hearing Scale (speech subscale). This subscale consists of 14 items and is scored on an 11-point visual analog scale.
fatigue | 1 day
  Fatigue will be measured with the Dutch ICF Activity Inventory (feeling fit subscale). This subscale consists of 9 items, scored on a 5-point likert scale. Secondly, the Fatigue Assessment Scale will be used, consisting of 10 items, scored on a 5-point likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth MA van Nispen, prof.dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
IPD cannot be shared if it includes identifiable information.